CLINICAL TRIAL: NCT03420833
Title: Metabolic Mapping and Cardiac Resynchronization (Aim 1)
Brief Title: Metabolic Mapping and Cardiac Resynchronization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong-Mei Cha (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, Yong-Mei Cha, Sponsor Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-003359; 1R01HL134864-01A1 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single-center, randomized cross-over study
Who Masked: Participant, Investigator
Masking Description: Participants randomly assigned to have CRT-ON or OFF. At 6 months, participant CRT function will be crossed over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CRT-On first, then CRT-Off (Experimental): Subjects will be randomized to have the cardiac resynchronization therapy pacemaker (CRT-P) programmed on in the first intervention period, and after six months the CRT function will be turned off in the second intervention period.
  Interventions: Device: Cardiac resynchronization therapy pacemaker (CRT-P)
- CRT-Off first, then CRT-On (Experimental): Subjects will be randomized to have the cardiac resynchronization therapy pacemaker (CRT-P) programmed off in the first intervention period, and after six months the CRT function will be turned on in the second intervention period.
  Interventions: Device: Cardiac resynchronization therapy pacemaker (CRT-P)

INTERVENTIONS:
Device: Cardiac resynchronization therapy pacemaker (CRT-P) — A pacemaker is an implantable, battery-powered minicomputer that sends electrical pulses to the heart whenever it detects a slow heartbeat or no heartbeat at all. When it senses a slow heartbeat or lack of heartbeat, it sends electrical impulses to restore a normal rhythm. Cardiac resynchronization therapy pacemakers, or CRT-Ps, treat heart failure by resynchronizing electrical impulses in the heart's four chambers, improving the heart's ability to pump blood to the body effectively and efficiently.
  Other Names: BIOTRONIK Evia HF-T

SUMMARY:
The purpose of this study is to gather information on the safety and effectiveness of cardiac resynchronization therapy (CRT) in patients who have mild heart failure (HF) and left bundle branch block (LBBB).

ELIGIBILITY:
Inclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) 35%-50%
* New York Heart Association (NYHA) class I-II
* QRS duration of ≥120ms
* Left bundle branch block (LBBB)
* Patient is able to receive a transvenous pectoral CRT implant
* Patient is able to sign informed consent
* Two echocardiograms are required to confirm a stable reduced LVEF
* Patient is on optimal and stable medical therapy (ACE inhibitor or angiotensin II type 1 (AT1 )blocker, beta blocker, etc. over the last 6 months)

Exclusion Criteria:

* Advanced comorbid conditions with life expectancy <1 year
* Patient is <18 of years of age
* Patient has a CRT device
* Female patients who is pregnant or not on a reliable form of birth control. Women of childbearing potential are required to have negative pregnancy test within the 7 days prior to device implant
* Unwilling or unable to return for required follow-up visits
* Patient decides study participation is cost-prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Mei Cha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 participants were enrolled, 6 withdrew prior study randomization.
Period: Overall Study
Arm/Group | CRT-On First, Then CRT-Off | CRT-Off First, Then CRT-On
Started | 38 | 38
Completed | 28 | 37
Not Completed | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT-On First, Then CRT-Off | CRT-Off First, Then CRT-On | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.8) | 68.3 (10.0) | 68.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 28 | 26 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 38 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricle End-Systolic Volume Index (LVESVI)
Description: LVESVI is the volume of blood in the left ventricle at the end of contraction, or systole, adjusted for the individual's body surface area.
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: mL/m^2
Groups:
- CRT-ON: Subjects who had their cardiac resynchronization therapy pacemaker (CRT-P) programmed ON in either the first six months or last six months of the study.
- CRT-OFF: Subjects who had their cardiac resynchronization therapy pacemaker (CRT-P) programmed OFF in either the first six months or last six months of the study.
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 72 | 66
mL/m^2 | -11.6 (12.8) | -4.1 (12.2)
Statistical Analysis 1: Comparison: CRT-ON; Test type: Superiority; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: CRT-OFF; Test type: Superiority; p = 0.009, t-test, 2 sided

2. Primary Outcome: Number of Subjects Experiencing Any System-Related Complications
Description: This is a composite endpoint; system-related complications could include any of the following: device pocket hematoma, pneumothorax, myocardial perforation, lead dislodgement, lead revision and device-related infection.
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 72 | 66
Participants | 2 | 2

3. Secondary Outcome: Number of Subjects Admitted to the Hospital for Heart Failure
Description: The total number of subjects hospitalized for heart failure during the study.
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Groups:
- CRT-OFF: Subjects who had their cardiac resynchronization therapy pacemaker (CRT-P) programmed ON in either the first six months or last six months of the study.
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 76 | 76
Participants | 0 | 0

4. Secondary Outcome: Change in N-Terminal Pro B-Type Natriuretic Peptide (NT-proBNP) by CRT Randomization From 6 Months to 12 Months
Description: The NT-proBNP is a substance that is produced in the heart and released when the heart is stretched and working hard to pump blood, measured in pg/mL. The change was calculated as the value at 12 months minus the value at 6 months.
Time Frame: 6 months, 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CRT-On First, Then CRT-Off | CRT-Off First, Then CRT-On
Number analyzed (Participants) | 27 | 32
pg/mL | 0.1 (0.6) | -0.3 (0.6)
Statistical Analysis 1: Comparison: CRT-On First, Then CRT-Off vs CRT-Off First, Then CRT-On; Test type: Superiority; p = 0.024, t-test, 2 sided

5. Secondary Outcome: Number of Subjects Who Experience Sustained Ventricular Tachycardia or Fibrillation Greater Than 30 Seconds
Description: In ventricular tachycardia, abnormal electrical signals in the ventricles cause the heart to beat faster than normal, usually 100 or more beats a minute, out of sync with the upper chambers. Ventricular fibrillation is the most serious cardiac rhythm disturbance. The lower chambers quiver and the heart can't pump any blood, causing cardiac arrest.
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 76 | 76
Participants | 1 | 0

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF)
Description: LVEF refers to how well your left ventricle (or right ventricle) pumps blood with each heart beat. Most times, EF refers to the amount of blood being pumped out of the left ventricle each time it contracts. The left ventricle is the heart's main pumping chamber.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 74 | 66
percent | 5.3 (8.2) | 2.2 (7.0)
Statistical Analysis 1: Comparison: CRT-ON; Test type: Superiority; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: CRT-OFF; Test type: Superiority; p = 0.011, t-test, 2 sided

7. Secondary Outcome: Number of Subjects Who Die in One Year
Description: The total number of subjects to die for any reason during the study.
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-ON | CRT-OFF
Number analyzed (Participants) | 76 | 76
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all participants from enrollment through the 48 month follow up visit, for a total of approximately 5 years.
Arm/Group | CRT-ON | CRT-OFF
All-Cause Mortality (participants affected / at risk) | 2/76 | 3/76
Serious Adverse Events (participants affected / at risk) | 6/76 | 8/76
Other Adverse Events (participants affected / at risk) | 44/76 | 29/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-ON (N=76) | CRT-OFF (N=76)
Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Lead dislodgment (General disorders) | 2 (2) | 0 (0)
Electrical Stimulation (General disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (General disorders) | 0 (0) | 3 (3)
Diaphragmatic Stimulation (General disorders) | 1 (1) | 0 (0)
Pneumothorax (General disorders) | 0 (0) | 1 (1)
Sepsis (General disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 0 (0) | 2 (2)
Ischemic Stroke (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-ON (N=76) | CRT-OFF (N=76)
Tenderness at implant site (General disorders) | 1 (1) | 0 (0)
Shortness of breath (General disorders) | 1 (1) | 1 (1)
Anemia (General disorders) | 11 (11) | 8 (8)
Hyperglycemia (General disorders) | 10 (10) | 10 (10)
Fatigue (General disorders) | 2 (2) | 2 (2)
Dizziness (General disorders) | 3 (3) | 2 (2)
COVID-19 (General disorders) | 3 (3) | 1 (1)
Dyspenea (General disorders) | 3 (3) | 2 (2)
Cough (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03420833/Prot_SAP_000.pdf